CLINICAL TRIAL: NCT05451641
Title: The Effect of Blood Flow Restriction Resistance Training on Vascular Function: Wide-Rigid Cuffs vs. Narrow-Elastic Bands
Brief Title: Blood Flow Restriction Resistance Training Intervention on Vascular Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00002999
Record Dates: First submitted 2022-06-22; First posted 2022-07-11 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Endothelial Function

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Wide-rigid cuff (Experimental): The wide-rigid cuff will be randomly assigned to one of the subject's arms.
  Interventions: Behavioral: Blood flow restriction resistance training
- Narrow-elastic band (Experimental): The narrow-elastic band will be randomly assigned to another arm of the subject.
  Interventions: Behavioral: Blood flow restriction resistance training

INTERVENTIONS:
Behavioral: Blood flow restriction resistance training — The participants will receive a 2-week exercise training program (3 times per week). Each training session will consist of 3 resistance training exercises with two blood flow restriction devices (wide-rigid cuff and narrow-elastic band). For both arms, the participants will perform the same exercise with different BFR devices.

SUMMARY:
The purpose of this study is to investigate the effect of blood flow restriction (BFR) resistance training on vascular function. The investigators aim to compare the effects of different BFR devices (wide-rigid cuffs and narrow elastic bands) on vascular function. The investigators hypothesize that BFR resistance training with wide-rigid cuffs might have a minor negative effect (short-term and reversible) on vascular function, while BFR resistance training with narrow-elastic bands may improve vascular function. Both training methods are equally effective in increasing muscle strength.

DETAILED DESCRIPTION:
Blood flow restriction (BFR) resistance training has been proven to be effective in increasing muscle mass and strength. During BFR training, cuffs (similar to blood pressure cuffs) are placed on the proximal ends of the extremities to partially occlude arterial blood flow to the working muscles and fully restrict venous outflow from the working muscle. The metabolites produced by the working muscle during exercise are trapped in the working muscle, which causes metabolic stress to augment muscle adaptation. Typically, two types of cuffs are used in the BFR training: the narrow-elastic bands and wide-rigid nylon cuffs adapted from surgical tourniquets and blood pressure cuffs.

Currently, the effect of BFR training on vascular function remains unclear. When the cuffs are removed after BFR training, there will be a reactive hyperemic blood flow to wash out all the metabolites produced during exercise. This reactive hyperemic blood flow also will impose shear stress on the arterial vessel wall. The shear stress will lead to an increase in vasodilator factors, which lead to an improvement in vascular function. However, other studies have pointed out that BFR training might cause a negative effect on vascular function when the occlusion pressure was too high. The possible mechanisms of the negative effect might be ischemia-reperfusion injury and retrograde shear stress in the artery. The wide-rigid cuffs are easily available but have the potential to inhibit the expansion of muscle upon increased blood flow accompanying exercise and muscle contraction while the narrow-elastic bands do not prevent the expansion. To the investigators' best knowledge, there is no study directly comparing different BFR cuffs on vascular function. Thus, the aim of the present study is to compare the effects of different BFR cuffs on vascular function (evaluated by flow-mediated dilation, a non-invasive measure of endothelial-derived vasodilation).

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy, sedentary or recreationally active young adults aged between 18 - 40 years old and signed the informed consent.

Exclusion Criteria:

* A current COVID-19 diagnosis
* morbid obesity
* hypertension
* smoking
* overt cardiovascular disease
* using any medication that might affect the cardiovascular system
* current participation in resistance training.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2022-09-20 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-19 (Actual)

PRIMARY OUTCOMES:
Change from baseline vascular function at 2 weeks | Baseline measurement and measurement at 2 weeks
  Flow-mediated dilation evaluated by an ultrasound machine
Change from baseline muscle strength at 2 weeks | Baseline measurement and measurement at 2 weeks
  Measured by a cable machine in the gym
Change from baseline grip strength at 2 weeks | Baseline measurement and measurement at 2 weeks
  Measured by a hand dynamometer

SECONDARY OUTCOMES:
Change from baseline body fat percentage at 2 weeks | Baseline measurement and measurement at 2 weeks
  Measured by a bioelectrical impedance analysis machine
Change from baseline fat mass at 2 weeks | Baseline measurement and measurement at 2 weeks
  Measured by a bioelectrical impedance analysis machine
Change from baseline lean body mass at 2 weeks | Baseline measurement and measurement at 2 weeks
  Measured by a bioelectrical impedance analysis machine
Blood flow responses to different types of cuff | Baseline measurement
  Measured by an ultrasound machine
Blood flow responses to different types of cuff | At 2 weeks
  Measured by an ultrasound machine
Change from baseline arterial stiffness at 2 weeks | Baseline measurement and measurement at 2 weeks
  Evaluated by the Omron VP-1000plus device (Non-invasive measurement)
Change from baseline blood lactate concentration | At 10 minutes before the training sessions (baseline measurement) and at 10 minutes after the training sessions
  Measured by a lactometer
Changes from baseline heart rate at the end of each exercise during all the training sessions | At 10 minutes before the training sessions (baseline measurement), at 10 minutes, 20 minutes, and 30 minutes during the training sessions
  Measured by a heart rate monitor
Change from baseline blood pressure at the end of each exercise during all the training sessions | At 10 minutes before the training sessions (baseline measurement), at 10 minutes, 20 minutes, and 30 minutes during the training sessions
  Measured by an Omron digital blood pressure monitor
Change of the perceived exertion | At 10 minutes, 20 minutes, and 30 minutes during the training sessions
  Borg rating of perceived exertion scale

CONTACTS AND LOCATIONS:
Overall Officials: Hirofumi Tanaka, PhD, Principal Investigator — The University of Texas at Austin
Locations (1):
- Cardiovascular Aging Research Laboratory, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lixandrao ME, Ugrinowitsch C, Berton R, Vechin FC, Conceicao MS, Damas F, Libardi CA, Roschel H. Magnitude of Muscle Strength and Mass Adaptations Between High-Load Resistance Training Versus Low-Load Resistance Training Associated with Blood-Flow Restriction: A Systematic Review and Meta-Analysis. Sports Med. 2018 Feb;48(2):361-378. doi: 10.1007/s40279-017-0795-y. PMID 29043659
- [Background] Pearson SJ, Hussain SR. A review on the mechanisms of blood-flow restriction resistance training-induced muscle hypertrophy. Sports Med. 2015 Feb;45(2):187-200. doi: 10.1007/s40279-014-0264-9. PMID 25249278
- [Background] Early KS, Rockhill M, Bryan A, Tyo B, Buuck D, McGinty J. EFFECT OF BLOOD FLOW RESTRICTION TRAINING ON MUSCULAR PERFORMANCE, PAIN AND VASCULAR FUNCTION. Int J Sports Phys Ther. 2020 Dec;15(6):892-900. doi: 10.26603/ijspt20200892. PMID 33344005
- [Background] Hunt JE, Galea D, Tufft G, Bunce D, Ferguson RA. Time course of regional vascular adaptations to low load resistance training with blood flow restriction. J Appl Physiol (1985). 2013 Aug 1;115(3):403-11. doi: 10.1152/japplphysiol.00040.2013. Epub 2013 May 23. PMID 23703116
- [Background] Horiuchi M, Okita K. Blood flow restricted exercise and vascular function. Int J Vasc Med. 2012;2012:543218. doi: 10.1155/2012/543218. Epub 2012 Oct 22. PMID 23133756
- [Background] Alhejily W, Aleksi A, Martin BJ, Anderson TJ. The effect of ischemia-reperfusion injury on measures of vascular function. Clin Hemorheol Microcirc. 2014;56(3):265-71. doi: 10.3233/CH-131741. PMID 23719421
- [Background] Thijssen DH, Dawson EA, Tinken TM, Cable NT, Green DJ. Retrograde flow and shear rate acutely impair endothelial function in humans. Hypertension. 2009 Jun;53(6):986-92. doi: 10.1161/HYPERTENSIONAHA.109.131508. Epub 2009 Apr 20. PMID 19380611